CLINICAL TRIAL: NCT03311698
Title: Homestead Agriculture and Nutrition Project in Rufiji District, Tanzania
Brief Title: Homestead Agriculture and Nutrition Project
Acronym: HANU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Ifakara Health Institute (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Chair, Department of Global Health and Population, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSPH-16-0397
Record Dates: First submitted 2017-09-27; First posted 2017-10-17 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Diet Modification; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Households receiving the intervention will receive (1) Interventions to promote homestead food production, increase agricultural production and food diversity, (2) nutritional counselling, including locally adapted instructions on the mix and quantity of food suitable for children of ages 6-24 months, and (3) a health-focused intervention, including information on micronutrient supplementation, integrated management of child illnesses, and prevention and management of child malnutrition with a focus on the first 1,000 days.
  Interventions: Behavioral: Nutrition-sensitive intervention
- Control (No Intervention): Households receive the standard of care in the area for agricultural and health services.

INTERVENTIONS:
Behavioral: Nutrition-sensitive intervention — Nutrition-sensitive intervention using behavior change communication on home gardening, diet, nutrition, WASH, and women's empowerment.
  Arms: Intervention

SUMMARY:
HANU is an evaluation of the effects of an integrated, gender-focused nutrition-sensitive intervention on the nutrition and health of young children and women of reproductive age in rural Tanzania.

DETAILED DESCRIPTION:
HANU aims to develop, implement, and evaluate nutrition-sensitive interventions among rural smallholder households in Rufiji Tanzania with the goal of improving the nutritional status and health of young children and women of reproductive age. Specifically, HANU will engage agricultural extension workers (AEWs) and community health workers (CHWs) to provide an integrated homestead food production, nutrition counselling, and public health intervention.

Households receiving the intervention will receive (1) Interventions to promote homestead food production, increase agricultural production and food diversity, (2) nutritional counselling, including locally adapted instructions on the mix and quantity of food suitable for children of ages 6-24 months, and (3) a health-focused intervention, including information on micronutrient supplementation, integrated management of child illnesses, and prevention and management of child malnutrition with a focus on the first 1,000 days. The intervention will include information on cultivation of nutrient-rich crop varieties, best practices for home gardening, safe water, sanitation, and hygiene practices (WASH), breastfeeding and complementary feeding, dietary intake and nutrition, and other basic public health messages. There are two delivery mechanisms for the intervention: farmer field schools and households visits. Household visits are conducted approximately bimonthly separately by AEWs and CHWs. Field schools are held approximately bimonthly and attended by both AEWs and CHWs. Households enrolled in the intervention will also receive agricultural inputs such as seeds, fertilizer, and watering cans.

Through this package of interventions, HANU aims to address the three primary pathways of impacting nutrition through agriculture: gender, income, and consumption. The interventions are designed to increase women's input into decision making over crop production and food consumption, child feeding, use of income, WASH practices, knowledge of nutrition and healthy diets; and home gardening skills. It also aims to address market barriers to homestead food production through connecting participants with agricultural services and helping to generate income through crop production.

The effects of the intervention will be evaluated through a cluster-randomized study design. Ten villages will be randomly selected and paired based on location, proximity to water, and population size. One village in each pair will be randomly assigned to receive the intervention (total of five villages) and one to the control group (total of five villages). Approximately 500 households in each arm will be screened, consented, and enrolled. Data will be collected by trained interviewers using surveys administered with electronic tablets at three time points, once at baseline, once 12 months after intervention implementation, and once approximately 36 months after intervention implementation. Anthropometric measurements of women and young children will be taken at three time points. Hemoglobin for women and young children will be measured among a subset of the study population at three time points.

Qualitative methods will be used to explore barriers to adopting the behaviors promoted through the intervention. One focus group discussion with study participants in each intervention village will be conducted to explore participant experiences with the interventions including key challenges. Eight key informant interviews will further assess sustainability aspects of the intervention.

It is possible that the adoption of home gardening practices and other positive nutrition and health behaviors could spillover to neighboring households. Therefore this study will also assess potential spillover effects of the intervention. In each intervention village, households that did not receive the intervention will be enrolled to assess potential spillover effects of the intervention through the use of a quantitative survey. Approximately 450 households will be enrolled and data will be collected at two time points 12 months after intervention implementation and 36 months after intervention implementation. One focus group discussion in each intervention village among households that did not receive the intervention will be conducted to further explore spillover effects.

ELIGIBILITY:
Households in one of the two study arms will be eligible for inclusion if they meet all of the following citeria:

* Provide informed consent
* Households with women of reproductive age and with at least one child under the age of 36 months (10 years for spillover households to ascertain the secondary outcomes of extent of spillover).
* Household has access to plot of land or containers where vegetables could be grown
* Households that speak and understand English or Swahili

Exclusion Criteria:

* Do not provide informed consent
* Households without a woman of reproductive age or a child under the age of 36 months (10 years for spillover households).
* Households without access to plot of land or containers where vegetables could be grown.
* Households that do not speak and understand English or Swahili.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participants must be a women of reproductive age
Enrollment: 1007 (Actual)
Dates: Start 2016-07-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Dietary diversity defined as number of food groups consumed out of 10 | 12 and 36 months
  Minimum dietary diversity for women of reproductive age defined as a minimum of 5 food groups consumed out of 10

SECONDARY OUTCOMES:
Child height/length | 12 and 36 months
  Height or length in centimeters
Child weight | 12 and 36 months
  Weight in kilograms
Child MUAC | 12 and 36 months
  Mid-upper arm circumference (MUAC) in centimeters
Women's Height | 12 and 36 months
  Height in centimeters
Women's weight | 12 and 36 months
  Weight in kilograms
Women's MUAC | 12 and 36 months
  Mid-upper arm circumference (MUAC) in centimeters
Hematologic status in women | 12 and 36 months
  hemoglobin (Hb) levels cut off points of Hb < 12 g/dl for non pregnant women and Hb < 11g/dl for pregnant women
Hematologic status in children | 12 and 36 months
  hemoglobin (Hb) levels cut off points of Hb < 11 g/dl
Child dietary diversity | 12 and 36 months
  Minimum dietary diversity for children under 4 years of age as defined by number of food groups consumed out of 10
Extent of spillover of home garden behavior | 12 and 36 months
  Has a home garden (binary)
Extent of spillover of vegetable crop production behavior | 12 and 36 months
  Number of vegetables grown in home garden
Extent of spillover of production and consumption of crops | 12 and 36 months
  Consumed vegetables grown in home garden (binary)
Early Childhood Development | 12 and 36 months
  Early Childhood Development (ECD) as measured by the Caregiver Reported Early Development Index (CREDI) using a continuous score of overall developmental status

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH); Honorati Masanja, PhD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Dar es Salaam, Mikocheni, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blakstad MM, Mosha D, Bellows AL, Canavan CR, Chen JT, Mlalama K, Noor RA, Kinabo J, Masanja H, Fawzi WW. Home gardening improves dietary diversity, a cluster-randomized controlled trial among Tanzanian women. Matern Child Nutr. 2021 Apr;17(2):e13096. doi: 10.1111/mcn.13096. Epub 2020 Nov 26. PMID 33241924
- [Derived] Mosha D, Canavan CR, Bellows AL, Blakstad MM, Noor RA, Masanja H, Kinabo J, Fawzi W. The impact of integrated nutrition-sensitive interventions on nutrition and health of children and women in rural Tanzania: study protocol for a cluster-randomized controlled trial. BMC Nutr. 2018 Sep 6;4:29. doi: 10.1186/s40795-018-0238-7. eCollection 2018. PMID 32153890